CLINICAL TRIAL: NCT07016178
Title: Innovative Cognitive Impairment Case Finding and Engagement for Diverse Participation in Alzheimer's Disease Care, Treatment, And Research
Acronym: INCLUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Nicole R. Fowler, PhD, Scientist, Indiana University Center for Aging Research, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25818
Record Dates: First submitted 2025-05-14; First posted 2025-06-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer Disease; Alzheimer's Disease (Incl Subtypes); Dementia; Cognitive Decline
Keywords: Brain Health Navigator; Passive Digital Marker (PDM); early detection; MCI; Alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDM+ (Experimental): Patients at participating clinics identified through the Passive Digital Marker (PDM) as at risk will be contacted for clinical follow up via Twistle, a secure text message platform prior to their next schedule primary care visit. Patients identified as at risk, PDM+, who confirm a cognitive concern via Twistle will be referred to the IU Health Brain Health Navigator (BHN), a clinical nurse embedded in primary care. . The BHN will deliver the IUH Brain Health Protocol to assess for reversible causes, initiate shared decision-making processes for care and treatment, assess for treatment eligibility, and complete a warm hand-off when appropriate. Additionally, the BHN will facilitate patient enrollment in the Indiana CTSI ALL IN research registry and/or the IU Biobank.
  Interventions: Behavioral: Acceptability and Feasibility of Twistle messaging for PDM+ patients

INTERVENTIONS:
Behavioral: Acceptability and Feasibility of Twistle messaging for PDM+ patients — PC patients identified by the PDM as high risk for developing or having undetected MCI or ADRD will receive the patient-informed message developed in Aim 2. The patient-informed message will include instructions for completing validated questions about subjective memory concerns. In addition, interested patients will have the option to schedule a visit with the BHN, or enroll in research opportunities.

SUMMARY:
Recent studies have highlighted the potential use of electronic health record (EHR) data for scalable and less biased identification of people who may have or be at risk of developing MCI or ADRD at the population level.8,9 Using data from the EHR in advance of PC visits can systematically identify patients with undetected MCI and ADRD. At Indiana University (IU), researchers developed a Passive Digital Marker (PDM) to enable early detection of ADRD with an 80% accuracy for one-year and three-year prediction horizons.8,9 Despite the accuracy of the PDM, the feasibility, acceptability, and overall effectiveness of its use for early detection of ADRD in PC remains unclear.

Building on this innovative tool and the ongoing engagement in IUH PC for early detection of ADRD, we propose a project to test the acceptability and feasibility of implementing the PDM in IUH PC to identify people with and at risk of MCI and ADRD and measure if we can increase patient engagement in research and evidence-based follow-up care with the IUH Brain Health Navigator (BHN). The BHN, is primary care based registered nurse with special training to conduct additional assessments of patients following a positive ADRD screen to identify possible underlying causes of cognitive impairment and assist the PCP to facilitate the patient's next steps for diagnostic assessment.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older; established patients of 12 selected clinics at IU Health PC who are identified by the PDM as high risk for developing or having undetected MCI or ADRD.

Exclusion Criteria:

* Patients younger than 65 years; new patients to IUH (less than 12 months); individuals whose primary language is neither English nor Spanish; and current diagnosis of ADRD or MCI.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3454 (Actual)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Implementation of the PDM to identify at risk patients | 3 months post index visit
  Implement the PDM, using IUH EHR data, to identify primary care patients aged 65 or older who a have undetected MCI or ADRD or who are at risk. Measured by the percentage of patients with subjective cognitive concerns, and their MoCA scores in comparison to match the epidemiological rates in the literature on undetected MCI and ADRD in PC (~11-60%).
2.1 Effectiveness of Patient-informed messaging | 3 months post index visit
  Evaluate the effectiveness of the patient-informed message using IUH's patient facing application, Twistle, in engaging PDM positive patients to complete a cognitive assessment with the BHN as measured by the percentage of patients who open the message.
2.2 Effectiveness of Patient-informed messaging | 3 months post index visit
  Evaluate the effectiveness of the patient-informed message using IUH's patient facing application, Twistle, in engaging PDM positive patients to complete a cognitive assessment with the BHN as measured by the percentage that engage with the message.
2.3 Effectiveness of Patient-informed messaging | 3 months post index visit
  Evaluate the effectiveness of the patient-informed message using IUH's patient facing application, Twistle, in engaging PDM positive patients to complete a cognitive assessment with the BHN as measured by the percentage of patients who answer the Subjective Cognitive Concerns questions.
2.4 Effectiveness of Patient-informed messaging | 3 months post index visit
  Evaluate the effectiveness of the patient-informed message using IUH's patient facing application, Twistle, in engaging PDM positive patients to complete a cognitive assessment with the BHN as measured by the percentage of patients who schedule a BHN appointment.

SECONDARY OUTCOMES:
Engage in clinical research | 3 months post index visit
  The BHN will screen patients for eligibility to participate in ADRD clinical trials and, with their consent, sign them up for the IU clinical research registry. Measured by the percentage of patients who consent to the IU CTSI All IN clinical research registry and/or the IU Biobank repository.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Fowler, PhD, Principal Investigator — Indiana University School of Medicine, and Regenstrief Institute; IU Center for Aging Research
Locations (1):
- IU Health Primary Care, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No